CLINICAL TRIAL: NCT01512511
Title: Prospective Randomized Trial Comparing Nitrous Oxide and Carbon Dioxide for Laparoscopic Cholecystectomy
Brief Title: Comparing Nitrous Oxide and Carbon Dioxide for Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahvaz Jundishapur University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mehdi Asgari, Principal Investigator, Ahvaz Jundishapur University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: u-89140
Record Dates: First submitted 2012-01-03; First posted 2012-01-19 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Pneumoperitoneum
Keywords: laparoscopic cholecystectomy; pneumoperitoneum; nitrous oxide; carbon dioxide
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nitrous oxide (Experimental): use nitrous oxide for pneumoperitoneum creation
  Interventions: Procedure: nitrous oxide use for pneumoperitoneum creation
- carbon dioxide (Placebo Comparator): use carbon dioxide for pneumoperitoneum creation
  Interventions: Procedure: nitrous oxide use for pneumoperitoneum creation

INTERVENTIONS:
Procedure: nitrous oxide use for pneumoperitoneum creation — use nitrous oxide for create pneumoperitoneum in laparoscopic cholecystectomy

SUMMARY:
There is no general agreement about the ideal gas for pneumoperitoneum. CO2, now in common use, has not compared to N2O sufficiently to disclose which one has minimal "physiological" invasiveness characters. Assigned randomly to carbon dioxide or nitrous oxide group, the hemodynamic and respiratory parameters (heart rate, mean arterial blood pressure, end-tidal CO2, minute ventilation, and O2 saturation) before pneumoperitoneum and during it were recorded. Pain, as perceived by patients, is measured 2, 4 and 24 hours after the procedure by visual analogue scale. Vomiting and use of analgesics and antiemetics were recorded and compared.

ELIGIBILITY:
Inclusion Criteria:

* developed gallstones
* candidates for laparoscopic cholecystectomy
* written informed consent
* ASA Score = 1&2

Exclusion Criteria:

* signs and complications of gallstones in admission include acute cholecystitis and suppurative cholangitis
* complete Inability to move
* severe physical or mental disorders leading to inability to communicate -Pregnancy and
* cancer

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
heart rate | At the start of laparoscopic surgery and Immediately after surgery.
  number of heartbeats per minute measured in At the start of laparoscopic surgery and Immediately after surgery.

SECONDARY OUTCOMES:
Mean arterial pressure | At the start of laparoscopic surgery and Immediately after surgery.
  average arterial pressure during a single cardiac cycle At the start of laparoscopic surgery and Immediately after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Asgari, PhD, Principal Investigator — Ahvaz Jundishapur University of Medical Sciences
Locations (1):
- Ahvaz jundishapur university of medical sciences; Razi Hospital, Ahvāz, Khuzestan, Iran